CLINICAL TRIAL: NCT04045470
Title: A Pilot of a Microdevice For In Situ Candidate Drug Screening in Cutaneous Lesions of T-Cell Lymphoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Cecilia Larocca, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-639
Record Dates: First submitted 2019-07-25; First posted 2019-08-05 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Cutaneous T Cell Lymphoma; Peripheral T Cell Lymphoma
Keywords: Cutaneous T Cell Lymphoma; Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Intervention Model Description: Expansion cohort may enroll only after initial cohort has completed enrollment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Initial Cohort (Experimental): * Patients with plaque or tumor skin lesions of cutaneous T cell lymphoma or peripheral T cell lymphoma
  * Mandatory skin biopsy for corollary studies will be obtained
  * Patients will undergo percutaneous placement of four total microdevice(s) into two skin lesions (2 MD per skin lesion)
  Interventions: Device: Microdevices; Other: Standard of care therapy
- Expansion Cohort (Experimental): * Only patients with plaque or tumor skin lesions of cutaneous T cell lymphoma or peripheral T cell lymphoma who plan to start systemic therapy as part of standard of care
  * Mandatory skin biopsy for corollary studies will be obtained
  * Patients will undergo percutaneous placement of four total microdevice(s) into two skin lesions (2 MD per skin lesion)
  * Participants will receive standard of care therapy and clinical course followed
  * Participants will undergo standard of care therapy as previously determined by treating oncologist and/or dermatologist prior to enrollment to study
  * Participants will not be assigned any treatment intervention
  Interventions: Device: Microdevices; Other: Standard of care systemic therapy

INTERVENTIONS:
Device: Microdevices — The microdevice was developed as a tool with the ultimate goal to help screen several existing and investigational drugs directly within a patient's tumor to identify what drugs are the most effective for treating a patient's cancer.
Other: Standard of care therapy — Participant to receive standard of care therapy as previously determined by participant's treating oncologist and/or dermatologist, which may include a skin-directed or systemic therapy
  Arms: Initial Cohort
Other: Standard of care systemic therapy — Participant to receive standard of care therapy as previously determined by participant's treating oncologist and/or dermatologist, which must include a systemic therapy.
  Arms: Expansion Cohort

SUMMARY:
This research is being done to study the safety of implanting and retrieving a microdevice that releases up to 19 drugs directly within a cancerous lesion as a possible tool to evaluate the effectiveness of several approved cancer drugs against cutaneous T cell lymphoma and peripheral T cell lymphoma

DETAILED DESCRIPTION:
This research study is a Pilot and Feasibility Study, which is the first time investigators are examining this study microdevice loaded with drugs in patients with cutaneous lesions of cutaneous T cell lymphoma (CTCL) or peripheral T cell lymphoma (PTCL) patients.

The FDA (the U.S. Food and Drug Administration) has not approved the use of all the drugs contained in the microdevice as a treatment for cutaneous or peripheral T cell lymphoma. All drugs used in this study are FDA approved. Some drugs are for different cancer indications. Romidepsin, vorinostat, bexarotene, brentuximab vedotin, pralatrexate, and mogamulizumab have been FDA approved for CTCL. The FDA has not approved the use of the microdevice as a tool to identify what cancer treatment is best for any disease.

In this research study, the investigators are investigating whether the microdevice loaded with 19 drugs can be safely inserted in and removed from cancerous skin lesion. The microdevice was developed as a tool with the ultimate goal to help screen several existing and investigational drugs directly within a patient's tumor to identify what drugs are the most effective for treating a patient's cancer.

This microdevice was investigated in laboratory studies and shown to help identify what drugs could be effective in treating a specific cancer type. The microdevice was able to release drugs only to the immediately surrounding tumor tissue in concentrations of one millionth of what is normally needed for a therapeutic dose. The microdevice can be retrieved along with a few millimeters of surrounding treated tumor tissue for analysis of tumor response to drug.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have clinical diagnosis of cutaneous T-cell lymphoma or peripheral T-cell lymphoma with cutaneous involvement supported by histological evaluation of skin lesions.
* Participants must have measurable cutaneous disease, based on the modified Severity Weighted Assessment Tool (mSWAT; definition provided in appendix E). Skin lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Two lesions are amenable to placement of multiple devices in terms of lesion size and location, as assessed by dermatologist (minimum diameter of 1.5 cm).
* Patient must have the following minimum washout period from previous treatments and cannot be on any systemic therapy at the time of implantation.

  * 2 week from topical therapies of lesional skin selected for implantation
  * 2 weeks from retinoids, interferons, vorinostat, romidepsin, therapeutic doses of oral corticosteroids (physiologic replacement doses of oral corticosteoids are allowed)
  * 4 weeks from phototherapy
  * 5 half-lives for systemic cytotoxic anticancer agents, monoclonal antibodies, and investigational therapy
  * 12 weeks from local radiation therapy of lesional skin selected for implantation
  * 15 weeks from systemic immunotherapy targeting PD-1/PD-L1
* Age minimum of age 18.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Participants will undergo laboratory testing within 28 days prior to the procedure. Participants must have marrow function as defined below:

  * absolute neutrophil count ≥500/mcL
  * platelets ≥50,000/mcL
* Participants must be evaluated by a dermatologist or medical oncologist who will determine the clinically appropriate treatment strategy based on clinical history and extent of disease. Systemic therapy will be mandatory for cohort 2/expansion cohort, not for cohort 1. Systemic therapy may be initiated anytime within 4 weeks of MD removal.
* Patients must be deemed medically stable to undergo percutaneous procedures by their treating cutaneous oncologist.
* Ability to understand and the willingness to sign a written informed consent document.
* Patients must be willing to undergo research-related genetic and transcriptomic sequencing (somatic and germline) and data management, including the deposition of de-identified genetic sequencing data in NIH central data repositories.
* Patient is considered to have capacity to properly follow instructions at home for the care of device(s) that will each have an attached thin guidewire protruding through the skin and fixed in place (see Appendix B).

Exclusion Criteria:

* Positive serum pregnancy test at screening visit.
* Uncorrectable bleeding or coagulation disorder known to cause increased risk with surgical or biopsy procedures
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in this study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who will receive standard of care systemic therapy are not allowed to start any new skin directed therapy (e.g. topical steroids, radiation, phototherapy) concurrent with first systemic therapy initiated after device implantation and retrieval. Should a patient clinically progress on first systemic therapy and require a change in treatment, skin directed therapies may be introduced.
* Patients unable to undergo treatment wash-out period due to rapidly progressive disease requiring immediate systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-12-11 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
To Quantify The Number Of Microdevice-Related Failures Or Adverse Events As Assessed By CTCAE v4.0 After Microdevice Placement and Removal | 2 years
  "Failure" will be considered any of the following:
  1. Any grade 3 or 4 adverse events associated with device placement or retrieval
  2. Any device resulting in "major" adverse events as listed below:
     * device unable to be found or unable to be retrieved
     * device invading into vessel or device embolism
     * infection or severe tissue damage or abnormal wound healing associated with device or procedure (as deemed by a neutral consultant e.g. dermatologist, ID specialist or surgeon)
     * severe allergic/hypersensitivity reaction
     * severe bleeding
  3. Any device resulting in *two or more* "minor" adverse events as listed below:
     * device migration more than 10 mm
     * device fracture not causing a major adverse event
     * mild allergic/hypersensitivity reaction
     * manageable pain associated with biopsy procedure
     * minor bleeding For purposes of this endpoint, safety will be evaluated on a per-patient level, where an event is defined as any "failure" observed among all implanted devices.
To Retrieve The Device With Sufficient Tissue Of Sufficient Quality | 2 years
  For the feasibility endpoint, a "successful" procedure will be defined as the ability to retrieve the device (by either skin punch biopsy tool or surgical excision) without damaging tumor tissue surrounding the microdevice to allow for immunohistochemistry analysis.
  For purposes of this endpoint, feasibility will be assessed on a per-device basis rather than a per-patient basis, with each device considered relatively independent in terms of placement, retrieval, and analysis.

SECONDARY OUTCOMES:
Local Intralesional Response To Clinically Relevant Cancer Agents In Cutaneous T Cell Lymphomas | 2 years
Intralesional Heterogeneity In Drug Response Using Quantitative Histopathologic Assessment Of Tumor Tissue | 2 years
  Comparison of tumor responses to like drug delivered from separate microdevices.
Assessment Of Microdevice-Predicted Tumor Response To Drug | 3 years
  Correlation of tumor response to drug released by microdevice compared with clinical response to systemic administration of like drug
Quantitative Assessment Of Drug Effect On The Tumor Microenvironment And Signal Pathways By Immunofluorescence | 5 years
  Descriptive statistics will be used to summarize the quantitative measurements in cell number of different immunophenotypes and quantify signal transduction cascades. Descriptive statistics will be employed to summarize the variance in different measures of drug-induced microenvironment changes across participants.
To Identify Genomic And Transcriptomic Biomarkers of Drug Response by Whole Exome and RNA Sequencing and Subsequent Correlations To Microdevice Predicted Tumor Response | 5 years
  Genetic alterations will be cataloged in terms of single nucleotide variants, insertions/deletions, and copy number changes and will be reported in a descriptive manner. Preliminary correlations between a specific genetic feature and specific clinical features will be tested using Fisher's exact test for categorical variables or the Wilcoxon Rank-Sum test for continuous variables. Analyses of correlations between genetic and clinical features in different specimen types and patient groups are exploratory, and will rely on descriptive statistics without formal hypothesis testing. For each genetic feature of interest (e.g. mutation, gene expression profile) we will divide patient samples into groups based on the presence or absence of the feature. We will then assess whether the presence of the feature is associated with clinical outcomes using odds ratios, or correlation between genetic feature and overall survival, using Kaplan Meier estimates, with 95% confidence intervals to each.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Larocca, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation